CLINICAL TRIAL: NCT00451659
Title: Characterization of Recently Deployed Veterans
Status: Completed | Type: Observational
Sponsor: Tuscaloosa Research & Education Advancement Corporation (Other)
Other Study IDs: 0053
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2007-03-23 (Estimated); Status verified 2007-03

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; Veterans; Deployed
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a retrospective chart review of recently deployed veterans who served during the Iraq conflicts and were seen at the TVAMC in the outpatient Primary Care outpatient clinic that was recently set-up for newly returning veterans since its inception through July 1, 2005. Identical data will be collected on non-combat veterans that were seen in other primary care clinics at the Tuscaloosa VA Medical Center during June 2004 and July 1, 2005. This information will be used for comparison with the Iraqi veterans group. The data will be retrieved from a computerized list of these patients. Charts will then be examined to determine sociodemographic, medical, psychiatric, and health care utilization characteristics.

DETAILED DESCRIPTION:
The information will also be used internally at the TVAMC to better define treatment needs and also used in presentations and possible publications at professional meetings and in journals.

While this study is designed to be hypothesis generating for large prospective studies, we hypothesize that a majority of the recently deployed veterans who served in the Iraq conflict are in need of basic primary health care needs for illnesses that are common place among patients within this age group, except for a higher than expected prevalence of mood and anxiety disorders compared to usual primary care treatment-seeking populations.

This study is a retrospective chart review of recently deployed veterans who served during the Iraq conflicts and were seen at the TVAMC in the outpatient Primary Care outpatient clinic that was recently set-up for newly returning veterans since its inception through July 1, 2005. Identical data will be collected on non-combat veterans that were seen in other primary care clinics at the Tuscaloosa VA Medical Center during June 2004 and July 1, 2005. This information will be used for comparison with the Iraqi veterans group. The data will be retrieved from a computerized list of these patients. Charts will then be examined to determine sociodemographic, medical, psychiatric, and health care utilization characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, any race or ethic origin, at least 19 years of age
* Patients must have been seen by a provider in the outpatient Primary Care Clinic that has recently been set-up to serve recently deployed veterans who served during the Iraq conflict

Exclusion Criteria:

* Patients who did not serve during the Iraq conflict

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2005-02; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori L Davis, MD, Principal Investigator — TVAMC
Locations (1):
- TVAMC, Tuscaloosa, Alabama, United States

REFERENCES:
- [Background] Wolfe J, Proctor SP, Erickson DJ, Heeren T, Friedman MJ, Huang MT, Sutker PB, Vasterling JJ, White RF. Relationship of psychiatric status to Gulf War veterans' health problems. Psychosom Med. 1999 Jul-Aug;61(4):532-40. doi: 10.1097/00006842-199907000-00018. PMID 10443762
- See also: Department of Veterans Affairs: VA War Related Illness and Injury Study Centers — http://www.va.gov/environagents